CLINICAL TRIAL: NCT01241838
Title: The Effect of Heart Rate on Cardiac Index in Patients With Left Ventricular Hypertrophy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient no of patients eligible for enrollment.
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 1717
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Left Ventricular Hypertrophy; Diastolic Dysfunction; Heart Failure; Heart Rate
Keywords: Heart failure; Left ventricular hypertrophy; Diastolic dysfunction
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal left ventricular size (Placebo Comparator): Postoperative patient with normal left ventricular size
  Interventions: Device: Pacemaker
- Left ventricular hypertrophy (Active Comparator): Postoperative patient with left ventricular hypertrophy
  Interventions: Device: Pacemaker

INTERVENTIONS:
Device: Pacemaker — Routine postoperative temporary pacemaker Rate change of 65-80-95-110-125 beats/second in random order at day 3-4 after operation

SUMMARY:
The purpose of this study is to compare the effect of heart rate on cardiac index in patients with or without left ventricular hypertrophy. The study will be conducted in postoperative heart surgery patients with a pacemaker.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled heart surgery including thoracotomy
* Ejection fraction > 45%
* Duration of QRS complex < 120 milliseconds
* Sinus rhythm
* Planned perioperative temporary pacemaker

Group: Left ventricular hypertrophy:

Thickness of interventricular septum and posterior wall >11 mm.

Group: No left ventricular hypertrophy:

Thickness of interventricular septum and posterior wall <11 mm.

Exclusion Criteria:

* Active endocarditis
* Severe mitral insufficiency
* No patient consent

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Cardiac index | At heart rates 65-80-95-110-125

SECONDARY OUTCOMES:
Mean arterial blood pressure | At heart rates 65-80-95-110-125
Ejection fraction | Heart rates of 65-80-95-110-120
  Echocardiographic index of systolic function
Strain | Heart rates of 65-80-95-110-125
  Echocardiographic index of systolic function
S-max | Heart rates of 65-80-95-110-125 beats per second
  Echocardiographic index of systolic function
E/E' | Heart rates of 65-80-95-110-125 beats per second
  Echocardiographic index of diastolic function
E/A ratio | Heart rates of 65-80-95-110-125 beats per second
  Echocardiographic index of diastolic function
E'/A' ratio | Heart rates of 65-80-95-110-125 beats per second
  Echocardiographic index of diastolic function
Isovolumetric relaxation index | Heart rates of 65-80-95-110-125 beats per second
  Echocardiographic index of diastolic function
IVRT/IVRT' | Heart rates of 65-80-95-110-125 beats per second
  Echocardiographic index of diastolic function
End diastolic volume | Heart rates of 65-80-95-110-125 beats per second
  Volume of left ventricle and end diastole
End systolic volume | Heart rates of 65-80-95-110-125 beats per second
  Volume of left ventricle at end systole

CONTACTS AND LOCATIONS:
Overall Officials: Peter Juhl-Olsen, M.D., Principal Investigator — Department of Anaesthesiology, Århus University Hospital
Locations (1):
- Department of Anaesthesiology, Århus University Hospital, Århus N, Denmark